CLINICAL TRIAL: NCT06531798
Title: Post-marketing Phase IV, Multicenter, Prospective Study to Observe the Safety and Tolerability of Breztri aerosphereTM Containing a Fixed Dose Combination of Budesonide 160 mcg/ Glycopyrronium 7.2 mcg/ Formoterol Fumarate Dehydrate 5 mcg in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Brief Title: Post-marketing Phase 4 Safety & Tolerability Study of Breztri aerosphereTM in Indian Patients With Chronic Obstructive Pulmonary Disease
Acronym: INDOS-B
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5980L00017
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Moderate to Severe COPD

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): It will be a single-arm interventional phase 4 clinical study where participants will receive treatment with Breztri aerosphereTM containing budesonide 160 mcg/ glycopyrronium 7.2 mcg/ formoterol fumarate dehydrate 5 mcg (Breztri aerosphereTM pMDI) two actuations twice daily through oral inhalation for 24 weeks.
  Interventions: Drug: Breztri Aerosphere

INTERVENTIONS:
Drug: Breztri Aerosphere — Budesonide 160 mcg/Glycopyrrolate 7.2 mcg/Formoterol fumarate dehydrate 5 mcg

SUMMARY:
The purpose of this study is to observe the safety and tolerability of Breztri aerosphereTM as maintenance treatment in Indian patients with moderate to severe COPD.

DETAILED DESCRIPTION:
Study details include:

The study duration will be 26 weeks The treatment duration will be 24 weeks

ELIGIBILITY:
Inclusion Criteria:

Patients with a physician-confirmed diagnosis of COPD

* With a history of one severe COPD exacerbation or two or more moderate COPD exacerbations in the preceding 12 months.
* Post-bronchodilator FEV1 should be between ≥30 % to <80% of the predicted normal.
* Both male and female patients are allowed in the study
* Female of Non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is 2 years post-menopausal)
* A urine pregnancy test must be negative at screening.
* female participant must follow effective contraceptive method as outlined in protocol
* Patients should be capable of giving signed informed consent

Exclusion Criteria:

* Significant diseases or conditions other than COPD, which, in the opinion of the Investigator, may put the subject at risk because of participation in the study or may influence either the results of the study or the subject's ability to participate in the study.
* Chest x-ray within 6 months before screening must be acceptable to the investigator. Subjects who have a chest x-ray that reveals clinically significant abnormalities not believed to be due to the presence of COPD should not be included. A chest x-ray must be conducted if the most recent chest x-ray is not available at the time of screening.
* Patients having moderate to severe exacerbations within 6 weeks before the Screening period.
* Female patients who are pregnant or lactating or planning a family during the study period.
* Patients with either a history of hypersensitivity to excipients of the study drug or drugs with a similar chemical structure or class to the study drug.
* Patients participating in any current or future interventional trial during the study will not be enrolled in the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
To observe the safety and tolerability of Breztri aerosphereTM as maintenance treatment in Indian patients with moderate to severe COPD | 24 weeks
  Percentage, nature, intensity, seriousness and causal relationship of AEs, SAEs, and AEs leading to discontinuation of study drug will be assessed